CLINICAL TRIAL: NCT05184322
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral Ecnoglutide Tablet in Healthy Adult Participants
Brief Title: XW004 To Evaluate the Safety, Tolerability, PK, and PD of Oral Ecnoglutide Tablet in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sciwind Biosciences APAC CO Pty. Ltd. (Industry)
Collaborators: Hangzhou Sciwind Biosciences Co., Ltd. (Industry); Sciwind Biosciences USA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW0503-1011
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a single centre, double-blind, randomised, multiple-dose, placebo-controlled study, including six cohorts (Cohorts 1A/1B, 2, 3, 4, 5, 6) with a semi-parallel design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1A/1B (Experimental): Cohort 1A/1B will enroll 14 healthy participants.
  Interventions: Drug: T2026; Drug: Placebo; Drug: Oral ecnoglutide tablet
- Cohort 2 (Experimental): Cohort 2 will enroll 14 healthy participants.
  Interventions: Drug: T2026; Drug: Placebo; Drug: Oral ecnoglutide tablet
- Cohort 3 (Experimental): Cohort 3 will enroll 14 healthy participants.
  Interventions: Drug: T2026; Drug: Placebo; Drug: Oral ecnoglutide tablet
- Cohort 4 (Experimental): Cohort 4 will enroll 14 otherwise healthy participants with obesity.
  Interventions: Drug: Oral ecnoglutide tablet; Drug: T2026; Drug: Placebo
- Cohort 5 (Experimental): Cohort 5 will enroll 14 otherwise healthy participants with obesity.
  Interventions: Drug: Oral ecnoglutide tablet; Drug: T2026; Drug: Placebo
- Cohort 6 (Experimental): Cohort 6 will enroll 14 otherwise healthy participants with obesity.
  Interventions: Drug: T2026; Drug: Oral ecnoglutide tablet

INTERVENTIONS:
Drug: T2026 — Once daily for 15 days.
  Other Names: Absorption enhancer excipient
  Arms: Cohort 1A/1B; Cohort 2; Cohort 3; Cohort 6
Drug: Placebo — Once daily for 15 days.
  Arms: Cohort 1A/1B; Cohort 2; Cohort 3
Drug: Oral ecnoglutide tablet — Once daily for 6 weeks.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 4
Drug: Oral ecnoglutide tablet — Once daily and titrated up in concentration to once every week during maintenance period.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 5
Drug: Oral ecnoglutide tablet — Once daily for 15 days.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 6
Drug: Oral ecnoglutide tablet — Once daily for 15 days.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 1A/1B
Drug: Oral ecnoglutide tablet — Once daily for 15 days.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 2
Drug: Oral ecnoglutide tablet — Once daily for 15 days.
  Other Names: GLP-1 analogue; XW004
  Arms: Cohort 3
Drug: T2026 — Once daily for 6 weeks.
  Other Names: Absorption enhancer excipient
  Arms: Cohort 4
Drug: Placebo — Once daily for 6 weeks.
  Arms: Cohort 4
Drug: T2026 — Once daily to once weekly for 12 weeks.
  Other Names: Absorption enhancer excipient
  Arms: Cohort 5
Drug: Placebo — Once daily to once weekly for 12 weeks.
  Arms: Cohort 5

SUMMARY:
XW004 is an acylated human glucagon-like peptide 1 (GLP-1) analogue and is being developed for type 2 diabetes mellitus (T2DM) and obesity management.

DETAILED DESCRIPTION:
This is a single centre, double-blind, randomised, multiple-dose, placebo-controlled study, including six cohorts (Cohorts 1A/1B, 2, 3, 4, 5, 6) with a semi-parallel design. The study is designed to evaluate the safety, tolerability, PK, and PD of oral ecnoglutide tablet in healthy participants. Participants will undergo a Screening period beginning up to 28 days (Cohort 1 to 4) and 42 days (Cohort 5 and 6 ) prior to randomisation/dose administration and will be required to sign an informed consent form (ICF) before undertaking any study specific procedures or assessments. Participants who meet all of the inclusion and none of the exclusion criteria will be enrolled. Eligible participants will be admitted to the CRU on Day -1 for review of inclusion and exclusion criteria prior to the start of study procedures on Day 1. A Safety Review Committee (SRC) will be established to monitor the progress of this trial and to make recommendations on whether to continue, modify or stop the trial for safety or ethical reasons.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female participants, aged 18 to 55 years (inclusive at the time of informed consenting);
* Participants must be in good general health, with no significant medical history, and have no clinically significant abnormalities on physical examination at Screening and/or before administration of study drug;
* Stable body weight for at least 3 months prior to Screening (i.e., <5% change) by self-declaration;
* Participants must have a Body Mass Index (BMI) ≥22.0 kg/m2 and <32.0 kg/m2 and weigh ≥55 kg at Screening (Cohorts 1A/1B to 3), or participants must have a BMI ≥30.0 kg/m2 and <40.0 kg/m2 and weigh ≥75 kg at Screening (Cohort 4, 5 and 6 only);

Key Exclusion Criteria:

* Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, may require treatment or render the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product (IP) or procedures or interfere with study assessments;
* Confirmed diagnosis of diabetes mellitus type 1, type 2, or of any other forms at any time, and/or occurrence of documented or suspected hypoglycaemic episodes within 12 months prior to Screening;
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Number and percentage of treatment emergent adverse events (TEAEs) and serious adverse events (SAE) | Up to 98 days
  Count of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Richard Friend, Principal Investigator — Nucleus Network Brisbane Clinic
Locations (1):
- Q-Pharm Pty Ltd (AKA Nucleus Network Brisbane), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No